CLINICAL TRIAL: NCT05131152
Title: Microvascular and Inflammatory Responses of 0.05 Cyclosporine Eye Drop (II) in Treatment of Mild to Moderate Dry Eye
Brief Title: Microvascular and Inflammatory Responses of 0.05 Cyclosporine Eye Drop (II) in Treatment of Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ186
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye
Keywords: dry eye; conjunctival micro-circulation; inflammation
MeSH Terms: conditions — Dry Eye Syndromes; Inflammation | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: The recruitment of subjects must meet the diagnosis criteria of DEWS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyclosporine group (Experimental): Mild DE patients: topical usage of 0.05% cyclosporine Eye Drops BID + 0.1% Sodium Hyaluronate Eye Drops QID, both use for 16 weeks.
  Moderate DE patients: topical usage of 0.05% cyclosporine Eye Drops BID +0.1% Sodium Hyaluronate Eye Drops QID, both use for 16 weeks, and 0.02% Fluoromethalone Eye Drops BID for 4 weeks.
  Interventions: Drug: Cyclosporine; Device: oculus keratograph, in vivo laser confocal microscopy, Functional slit lamp biomicroscopy
- control group (Experimental): Mild DE patients: 0.1% Sodium Hyaluronate Eye Drops QID for 16 weeks Moderate DE patients: 0.02% Fluoromethalone Eye Drops BID for 4 weeks +0.1% Sodium Hyaluronate Eye Drops QID for 16 weeks.
  Interventions: Device: oculus keratograph, in vivo laser confocal microscopy, Functional slit lamp biomicroscopy

INTERVENTIONS:
Drug: Cyclosporine — 0.05% cyclosporine Eye Drops; Sodium Hyaluronate Eye Drops, 0.02% Fluoromethalone Eye Drops.
  Arms: cyclosporine group
Device: oculus keratograph, in vivo laser confocal microscopy, Functional slit lamp biomicroscopy — oculus keratograph, in vivo laser confocal microscopy, Functional slit lamp biomicroscopy

SUMMARY:
To explore the law of changes in ocular surface inflammation when 0.05% cyclosporine eye drops (II) is used to treat dry eye, 50 cases of mild to moderate dry eyes were included. The expectation is finding out whether cyclosporine has a regulatory effect on conjunctival microvascular parameters and other inflammation indicators after cyclosporine eye drops treat dry eye, and analyze the value of conjunctival microvascular indicators in dry eye immunosuppressive therapy.

DETAILED DESCRIPTION:
Dry eye is a common ocular surface disease that affects people's visual function and quality of life. In recent years, with the changes of lifestyles, the prevalence of dry eye is gradually increased. According to the consensus definition of Chinese dry eye experts in 2020, dry eye is a chronic ocular surface disease caused by multiple factors, while inflammation is emphasized as an important role in the occurrence and development of dry eye. Therefore, in addition to use artificial tears to alleviate the symptoms of dry eye, it is clinically recommended to combine low-concentration ocular surface hormones or immunosuppressant for anti-inflammatory therapy. As an immunosuppressant, cyclosporine can inhibit the infiltration of CD4+ T cells on the ocular surface, inhibit the apoptosis of conjunctival goblet and lacrimal gland acinar cells, and effectively alleviate ocular surface inflammation. In addition, cyclosporine can inhibit the calcineurin pathway by forming an intracellular complex with cyclophilin, promote the production of tears, and increase the density of goblet cells. Cyclosporine has an impact on many molecules in the immune pathway of dry eye.

However, how to use and adjust immunosuppressant according to the ocular surface inflammation still depends on the subjective experience of doctors, and there is no uniform standard. Therefore, finding biological reference indicators for ocular surface inflammation is the key to promoting the standardization and precision of anti-inflammatory drugs. The stimulation of inflammation factors can lead to the expansion of the capillary network, thus, the function of ocular surface capillaries can be used as an important indicator of ocular surface inflammation. Now, the intelligent analysis technology based on ocular surface micro vessels owned by my research team can clearly obtain blood flow imagines and topographic maps of blood vessel distribution in conjunctival micro vessels, and quantify the changes in microvascular shape, density and complexity, which is a kind of non-contact and convenient evaluation method. In our previous studies, it was confirmed that the treatment of moderate to severe dry eye with low concentrations of ocular surface hormones can cause changes of ocular surface microvascular parameters. Investigators hope to further observe the temporal and spatial changes of ocular surface microvascular function during the treatment of dry eye with cyclosporine, and correlation with inflammatory cells, inflammatory factors and neuroinflammation, explore the effect of the drug on dry eye related inflammation target issues and the guiding value of conjunctival microvascular indicators in dry eye immunosuppressive therapy, in order to change the previous dry eye anti-inflammatory treatment and the mode of medication based on the doctor's personal experience.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* meet the 2-3 grade dry eye diagnosis: 1) At least one eye has one or more ocular discomfort symptoms and OSDI score ≥23; 2) At least one eye meets one of the following two: 2 mm/5min≤Schirmer I test (no anesthesia) <10 mm/5min; BUT≤10s. 3) Corneal spotting but no extensive erosion.

Exclusion Criteria:

* Contact lens wearers;
* Allergies to the study drug;
* Active eye infections; history of serious systemic diseases;
* Pregnancy or breastfeeding;
* Receiving or starting other treatments that may interfere with the interpretation of the results;
* Participating any other clinical trials within 3 months;
* Previous eye surgery, including laser treatment and refractive surgery;
* Need or have undergone punctal embolization or nasolacrimal duct obstruction;
* KCS secondary to the destruction of conjunctival goblet cells (such as vitamin A deficiency) ;
* Scar formation (such as cicatricial pemphigus, alkali burn, trachoma or radiation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Conjunctival microvascular blood flow velocity | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  Achieved by Functional slit lamp Biomicroscopy: a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital. camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.

SECONDARY OUTCOMES:
Tear collection and analysis | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  After communicating with the patient, 5 μL of tear fluid was collected with a 5 μL capillary tear collector at the medial and lateral canthus (collected three times per eye and mixed the tears from the left and right eyes into one centrifuge tube). The sample was transferred into Centrifuge tubes and stored at -80 °C until further analysis. Cytokine concentrations were measured using microsphere-based immunoassay analysis.

OTHER OUTCOMES:
Conjunctival microvascular blood flow | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
Df (vascular complexity index) | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
D0 (vascular density index) | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
Conjunctival microvascular diameter | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
The hyperemia index | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  The hyperemia index (HI) was measured by determining the percentage of conjunctival microvascular area in the conjunctiva automatically. The subjects were required to keep their eyes open and focus on the illuminated ring in front. Three consecutive readings were recorded, and the median was used. All data were recorded and analyzed with TF-scan software in the system of Keratograph 5M (Oculus, Wetzlar, Germany).
Ocular Surface Disease Index (OSDI) | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  The dry eye diagnosis flowchart begins with history-taking, risk factors are questioned in suspicious cases, and a screening test such as the Ocular Surface Disease Index (OSDI) Questionnaire is applied.
Non-invasive tear-film break-up time | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  Non-invasived tear-film break-up time is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) with a scale of seconds. Higher values represent a better outcome.
Schirmer I test | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  The tear production was measured with Schirmer strips without anaesthesia 15 minutes after corneal staining.
Corneal Fluorescein Staining | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale (0-3 scale for each area of 5 areas, total score 15). Higher values represent a worse outcome.
Infrared imaging of meibomian gland | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  Infrared photography of the upper meibomian glands were measured and imaged by tear film and meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany).
In Vivo Confocal imaging | 12 weeks after commencement of treatment-16 weeks after commencement of treatment
  IVCM image acquisition for all DE patients was completed using the in vivo corneal confocal microscopy (Heidelberg Engineering GmbH, 101 Heidelberg, Germany).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China